CLINICAL TRIAL: NCT02192359
Title: A Phase I Study of Intracranially Administered Carboxylesterase-Expressing Neural Stem Cells in Combination With Intravenous Irinotecan in Patients With Recurrent High-Grade Gliomas
Brief Title: Carboxylesterase-Expressing Allogeneic Neural Stem Cells and Irinotecan Hydrochloride in Treating Patients With Recurrent High-Grade Gliomas
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14108; NCI-2014-01463 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14108 (Other: City of Hope Medical Center); P30CA033572 (NIH); R01CA198076 (NIH)
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Results first posted 2024-04-29 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Anaplastic Astrocytoma; Recurrent Anaplastic Oligoastrocytoma; Recurrent Anaplastic Oligodendroglioma; Recurrent Glioblastoma; Recurrent Gliosarcoma; Recurrent Malignant Glioma; Recurrent WHO Grade III Glioma
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Glioma | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (hCE1m6-NSCs and irinotecan hydrochloride) (Experimental): Patients receive carboxylesterase-expressing allogeneic neural stem cells intracranially over 1.5-4.5 hours on days 1 and 15 (day 1 only for patients at dose level 1) and irinotecan hydrochloride IV over 90 minutes on days 3 and 17. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Carboxylesterase-expressing Allogeneic Neural Stem Cells; Drug: Irinotecan; Drug: Irinotecan Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Carboxylesterase-expressing Allogeneic Neural Stem Cells — Given intracranially
  Other Names: CE-secreting Allogeneic NSCs; hCE1m6-NSC
Drug: Irinotecan — Given IV
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; U-101440E; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of carboxylesterase-expressing allogeneic neural stem cells when given together with irinotecan hydrochloride in treating patients with high-grade gliomas that have come back. Placing genetically modified neural stem cells into brain tumor cells may make the tumor more sensitive to irinotecan hydrochloride. Irinotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving carboxylesterase-expressing allogeneic neural stem cells and irinotecan hydrochloride may be a better treatment for high-grade gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To define the recommended phase II doses (RP2D) of intracranially administered carboxylesterase-expressing allogeneic neural stem cells (hCE1m6-NSCs) in combination with intravenous irinotecan in patients with recurrent high grade glioma.

SECONDARY OBJECTIVES:

I. To describe the relationship between hCE1m6-NSC dose and SN-38 (SN-38) concentrations in brain interstitium.

II. To characterize the relationship between intracerebral and systemic concentrations of irinotecan (irinotecan hydrochloride) and SN-38.

III. To investigate the biologic activity of hCE1m6 NSCs by comparing SN-38 concentrations in the brain after treatment with hCE1m6-NSCs and irinotecan versus irinotecan alone.

IV. To assess for possible development of adenovirally transduced neural stem cell (NSC) immunogenicity after first exposure and with repeat doses of NSCs.

V. To describe the clinical benefit (defined as stable disease, partial response, or complete response) in patients who receive treatment with repeat cycles of NSCs and irinotecan.

VI. To determine, at time of autopsy, the fate of the NSCs.

OUTLINE: This is a dose-escalation study of carboxylesterase-expressing allogeneic neural stem cells.

Patients receive carboxylesterase-expressing allogeneic neural stem cells intracranially over 1.5-4.5 hours on days 1 and 15 (day 1 only for patients at dose level 1) and irinotecan hydrochloride intravenously (IV) over 90 minutes on days 3 and 17. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 3 and 6 months, and then annually thereafter for a minimum of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be able to understand and be willing to sign a written informed consent document
* Participant must be willing to comply with study and/or follow-up procedures
* Karnofsky performance status >= 70%
* Life expectancy of >= 3 months
* Histologically-confirmed diagnosis of a grade III or IV glioma (including glioblastoma, anaplastic astrocytoma, gliosarcoma, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma), or has a prior, histologically-confirmed, diagnosis of a grade II glioma and now has radiographic findings consistent with a high-grade glioma (grade III or IV)
* Imaging studies show evidence of recurrent tumor(s); if a patient is going to be enrolled to dose level two or higher, the patient must have a component of supratentorial disease (so as to enable placement of a Rickham reservoir/catheter) that is amenable to resection or biopsy
* High-grade glioma has recurred or progressed after prior treatment with brain radiation and temozolomide
* Participant must be in need of a craniotomy for tumor resection or a stereotactic brain biopsy for the purpose of diagnosis or differentiating between tumor progression versus treatment-induced effects following radiation therapy +/- chemotherapy
* Based on the neurosurgeon?s judgment, there is no anticipated physical connection between the post-resection tumor cavity and the cerebral ventricles
* Neurosurgeon finds the prospective participant is able to undergo neurosurgery
* Any number of prior therapies is permitted; from the start of study treatment, the following time periods must have elapsed: 6 weeks from nitrosourea-containing chemotherapy, 4 weeks from non-nitrosourea-containing cytotoxic chemotherapy (except 23 days from last daily dose of temozolomide taken in a 5 of 28 day regimen), and 2 weeks from last dose of a targeted agent (except 4 weeks for bevacizumab); there is no time period requirement for prior radiation therapy
* Any clinically significant toxicity from prior therapy must have improved to grade 0 or grade 1
* Absolute neutrophil count (ANC) >= 1,500 cells/ul
* Platelets > 100,000 cells/ul
* Total bilirubin =< 2.0 mg/dl
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 4 times institutional upper limit of normal
* Serum creatinine =< 1.5 x the institutional upper limit of normal
* Homozygous negative for the UDP glucuronosyltransferase 1 family, polypeptide A1 (UGT 1A1)*28 allele
* Absence anti-human leukocyte antigen (HLA) antibodies specific for HLA class I antigens expressed by the coagulation factor III (thromboplastin, tissue factor) (F3).cytosine deaminase (CD).carboxylesterase (CE) NSCs
* Negative serum pregnancy test (women of childbearing potential only)
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception while participating in this study; women of childbearing potential must have a negative pregnancy test < 2 weeks prior to registration

Exclusion Criteria:

* Prior therapy with neural stem cells
* Use of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers including hepatic enzyme-inducing anticonvulsants (phenytoin, fosphenytoin, carbamazepine, phenobarbital, primidone, oxcarbazepine) within 2 weeks prior to start of study treatment
* Use of moderate to strong CYP3A4 inhibitors within 2 weeks prior to start of study treatment
* Use of drugs known to inhibit UGT1A1, such as atazanir, gemfibrozil, indinavir, or ketoconazole, within 2 weeks prior to start of study treatment
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids, such as systemic cyclosporine and tacrolimus; consult principal investigator for questions, including necessary washout period for the specific drug
* Flucytosine within 2 weeks prior to start of study treatment
* Use of herbal medications
* Current use (or planned use during the treatment period) of other investigational agents, or biological, chemotherapy, radiation or other anti-tumor therapy
* Patient has known human immunodeficiency virus (HIV) or hepatitis C infection; baseline testing for HIV or hepatitis C is not required
* Prospective participant is unable to undergo a magnetic resonance imaging (MRI) with contrast agent
* Known chronic or active viral infections of the central nervous system (CNS)
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Diagnosis of Gilbert?s disease
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan
* Known sensitivity to any of the products to be administered during dosing
* Any other active malignancy
* Pregnant women and women who are lactating
* Serious medical or psychiatric illness that could, in the investigator?s opinion, potentially interfere with the safety monitoring requirements and completion of treatment according to this protocol
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2026-09-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jana L Portnow, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: 5x10^7 (1 Dose): Carboxylesterase-expressing Allogeneic Neural Stem Cells: Given intracranially, 5x10^7 (1 dose)
  Irinotecan: 180 mg/m2
- Dose Level 2: 5x10^7 (2 Doses): Carboxylesterase-expressing Allogeneic Neural Stem Cells: Given intracranially, 5x10^7 (2 doses)
  Irinotecan: 180 mg/m2
- Dose Level 3: 1x10^8 (2 Doses): Carboxylesterase-expressing Allogeneic Neural Stem Cells: Given intracranially, 1x10^8 (2 doses)
  Irinotecan: 180 mg/m2
- Dose Level 4: 1.5x10^8 (2 Doses): Carboxylesterase-expressing Allogeneic Neural Stem Cells: Given intracranially, 1.5x10^8 (2 doses)
  Irinotecan: 180 mg/m2
Period: Overall Study
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 3: 1x10^8 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
Started | 4 | 3 | 4 | 7
Completed | 3 | 3 | 3 | 6
Not Completed | 1 | 0 | 1 | 1
Not completed — Taken off study treatment due to persistent gr 2 decreased platelets requiring transfusions | 0 | 0 | 1 | 0
Not completed — Could not receive irinotecan due to low KPS score post surgery | 1 | 0 | 0 | 0
Not completed — Taken off study treatment to catheter infection not related to treatment | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 3: 1x10^8 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses) | Total
Number analyzed (Participants) | 4 | 3 | 4 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 6 | 17
  >=65 years | 0 | 0 | 0 | 1 | 1
Age, Continuous [Median (Full Range); unit: years] | 49.5 [25 to 58] | 56 [55 to 57] | 56.5 [32 to 62] | 44 [32 to 65] | 51 [25 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 0 | 3
  Male | 4 | 1 | 3 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 3 | 4 | 9
  Not Hispanic or Latino | 3 | 2 | 1 | 3 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 2 | 4 | 7 | 17
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 4 | 7 | 18
Tumor Type [Count of Participants; unit: Participants]
  anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligoastrocytoma | 1 | 0 | 1 | 2 | 4
  glioblastoma, gliosarcoma | 3 | 3 | 3 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose-limiting Toxicity (DLT)
Description: Toxicities will be graded using NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. A DLT is defined as an adverse event that is related to the administration of NSCs and/or irinotecan, occurs during the first treatment cycle and meets any of the following:
  1. Received less than 80% of study treatments except due to CNS toxicity
  2. Grade 4 thrombocytopenia or anemia or neutropenia lasting > 7 days
  3. Febrile neutropenia with ANC < 0.5 x10^9/L
  4. Grade 3 central nervous system (CNS) disorder lasting > 7 days not attributed to tumor or surgery and not present at baseline
  5. Second occurrence of grade 3 CNS disorder not attributed to tumor or surgery and not present at baseline
  6. Any grade 4 CNS disorder not attributed to tumor or surgery and not present at baseline
  7. Grade 3 toxicity despite therapy lasting > 7 days
  8. Grade 3 toxicity resulting in study agent discontinuation
  9. Grade 4 toxicity, except grade 4 diarrhea responding to therapy within 3 days
Time Frame: 28 days post first dose of NSC treatment on day 1, cycle 1
Population: 1 participant in each of dose levels 1, 3, and 4 was not evaluable for DLT because they were removed from the study due to adverse events not related to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 3: 1x10^8 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
Number analyzed (Participants) | 3 | 3 | 3 | 6
Participants | 0 | 0 | 0 | 1

2. Primary Outcome: Number of Participants With Grade 3 or Higher Toxicity Profile Attributed to NSCs
Description: Grade 3 or higher toxicity profile as assessed by the NCI CTCAE version version 4.0. Toxicities reported are possibly, probably or definitely related to NSCs.
Time Frame: Followed 30 days post treatment for all toxicities (min=33,max 142 days), up to 5 years for gene therapy toxicities
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 3: 1x10^8 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
Number analyzed (Participants) | 4 | 3 | 4 | 7
Participants | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Grade 3 or Higher Toxicity Profile Attributed to Irinotecan
Description: Grade 3 or higher toxicity profile as assessed by the NCI CTCAE version version 4.0. Toxicities reported are possibly, probably or definitely related to Irinotecan.
Time Frame: Followed 30 days post treatment for all toxicities (min=33,max 142 days), up to 5 years for gene therapy toxicities
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 3: 1x10^8 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
Number analyzed (Participants) | 4 | 3 | 4 | 7
Participants
  Fatigue: Yes | 0 | 0 | 1 | 0
  Fatigue: No | 4 | 3 | 3 | 7
  Platelet count decreased: Yes | 1 | 0 | 0 | 0
  Platelet count decreased: No | 3 | 3 | 4 | 7
  White blood cell decreased: Yes | 1 | 0 | 0 | 0
  White blood cell decreased: No | 3 | 3 | 4 | 7
  Meningitis: Yes | 0 | 1 | 0 | 0
  Meningitis: No | 4 | 2 | 4 | 7
  Hypophosphatemia: Yes | 0 | 1 | 0 | 0
  Hypophosphatemia: No | 4 | 2 | 4 | 7
  Brain abscess: Yes | 0 | 0 | 1 | 0
  Brain abscess: No | 4 | 3 | 3 | 7
  Catheter related infection: Yes | 0 | 0 | 0 | 1
  Catheter related infection: No | 4 | 3 | 4 | 6

4. Secondary Outcome: Median Ratio of SN-38 Area Under the Curve (AUC) to CPT-11 AUC in Plasma
Description: Pharmacokinetic data from patients who undergo intracerebral microdialysis will be summarized using descriptive statistics. hCE1m6-NSC dose and liposomal SN-38 concentrations in brain interstitium using microdialysis data from the patients treated with the initial neural stem cells (NSC) doses and from the patients in the cohort treated with the highest NSC dose. Ratios are reported as ratio x 100.
Time Frame: Pre-dose, at 90 minutes (just prior to the end of the infusion), and then at 30 minutes, 1, 2, 4, 8, 24, and 48 hours after the end of the infusion after day 1, cycle 1
Population: All 4 participants in dose level 3 and one participant in dose level 4 did not have plasma samples collected.
Measure: Median (Full Range); unit: ratio x 100
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
Number analyzed (Participants) | 3 | 3 | 6
ratio x 100 | 4.8 [3.8 to 5.5] | 0.8 [0.3 to 1.7] | 2.35 [1.2 to 3.8]

5. Secondary Outcome: Median Ratio of SN-38 AUC to CPT-11 AUC in the Brain
Description: Pharmacokinetic data from patients who undergo intracerebral microdialysis will be summarized using descriptive statistics. hCE1m6-NSC dose and liposomal SN-38 concentrations in brain interstitium using microdialysis data from the patients treated with the initial neural stem cells (NSC) doses and from the patients in the cohort treated with the highest NSC dose. Ratio is reported as ratio x 100
Time Frame: as for outcome 4
Population: All 4 participants in dose level 3 did not have brain samples collected.
Measure: Median (Full Range); unit: ratio x 100
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
Number analyzed (Participants) | 3 | 3 | 7
ratio x 100 | 6.9 [6.0 to 9.3] | 8.8 [4.9 to 28.2] | 12.2 [3.7 to 26.3]

6. Secondary Outcome: Number of Participants With Clinical Benefit Defined by Response Assessment in Neuro-Oncology (RANO)
Description: Clinical benefit is defined by participants achieving stable disease (SD), partial response (PR), or complete response (CR).
  CR: Complete disappearance of all enhancing disease (measurable and nonmeasureable) that is sustained for at least 4 weeks, stable or improved non-enhancing FLAIR/T2 lesions, no new lesions, off corticosteroids (physiologic replacement doses allowed), and neurologically stable or improved.
  PR: ≥ 50% decrease of all measurable enhancing lesions, sustained for at least 4 weeks, no progression of non-measurable disease, stable or improved non-enhancing FLAIR/T2 lesions, no new lesions, corticosteroid dose stable or reduced (compared to baseline), and neurologically stable or improved.
  SD: Does not qualify for CR, PR, or PD, stable non-enhancing FLAIR/T2 lesions, stable or reduced corticosteroids (compared to baseline), clinically stable.
Time Frame: Until death or disease progression, a median of 2 months, up to 6 months
Population: 1 participant in dose levels 1 and 3 and 2 is dose level 4 were unevaluable for response due to not receiving the full treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 3: 1x10^8 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
Number analyzed (Participants) | 3 | 3 | 3 | 5
Participants | 0 | 1 | 1 | 3

ADVERSE EVENTS:
Time Frame: Followed 30 days post treatment for all toxicities (min=33,max 142 days) up to 5 years for gene therapy toxicities
Arm/Group | Dose Level 1: 5x10^7 (1 Dose) | Dose Level 2: 5x10^7 (2 Doses) | Dose Level 3: 1x10^8 (2 Doses) | Dose Level 4: 1.5x10^8 (2 Doses)
All-Cause Mortality (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 6/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3 | 2/4 | 5/7
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: 5x10^7 (1 Dose) (N=4) | Dose Level 2: 5x10^7 (2 Doses) (N=3) | Dose Level 3: 1x10^8 (2 Doses) (N=4) | Dose Level 4: 1.5x10^8 (2 Doses) (N=7)
Brain abscess (Infections and infestations) | 0 | 0 | 1 | 0
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 0 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Altered mental status (Nervous system disorders) | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1: 5x10^7 (1 Dose) (N=4) | Dose Level 2: 5x10^7 (2 Doses) (N=3) | Dose Level 3: 1x10^8 (2 Doses) (N=4) | Dose Level 4: 1.5x10^8 (2 Doses) (N=7)
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 3 | 4
Sinus bradycardia (Cardiac disorders) | 2 | 2 | 0 | 5
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 3 | 3
tachypnea (Cardiac disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 1
Blurred vision (Eye disorders) | 1 | 0 | 1 | 1
Photophobia (Eye disorders) | 1 | 0 | 0 | 0
limited peripheral vision (Eye disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Bloating (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 3 | 5
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2
dry throat (Gastrointestinal disorders) | 0 | 0 | 1 | 0
thrush (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Edema face (General disorders) | 0 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 3
Fatigue (General disorders) | 3 | 2 | 3 | 6
Fever (General disorders) | 0 | 0 | 1 | 2
Gait disturbance (General disorders) | 0 | 1 | 4 | 3
Irritability (General disorders) | 0 | 0 | 1 | 3
Pain (General disorders) | 1 | 3 | 4 | 3
Edema limbs (General disorders) | 2 | 1 | 2 | 2
Localized edema (General disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
balance impairment (General disorders) | 0 | 0 | 1 | 0
generalized weakness (General disorders) | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Intraoperative head and neck injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Leakage from microdialysis catheters (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 1 | 3
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increase (Investigations) | 1 | 1 | 1 | 1
Lymphocyte count decreased (Investigations) | 3 | 2 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1 | 2 | 1
Platelet count decreased (Investigations) | 1 | 2 | 1 | 1
Weight loss (Investigations) | 2 | 0 | 1 | 0
White blood cell decreased (Investigations) | 1 | 2 | 2 | 0
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 2 | 3 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 2 | 3 | 3 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 2
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Joint range of motion decreased ce (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Right upper extremity twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Aphonia (Nervous system disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 1 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 1 | 2
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 1
Concentration impairment (Nervous system disorders) | 0 | 1 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2
Dysarthria (Nervous system disorders) | 2 | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Dysphasia (Nervous system disorders) | 1 | 1 | 1 | 3
Headache (Nervous system disorders) | 3 | 2 | 4 | 7
Hypersomnia (Nervous system disorders) | 2 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 2
Seizure (Nervous system disorders) | 2 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 2 | 1 | 0 | 2
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 1 | 2 | 1
balance impairment (Nervous system disorders) | 0 | 1 | 0 | 0
facial twitching (Nervous system disorders) | 0 | 1 | 0 | 0
pseudomeningocele (Nervous system disorders) | 0 | 1 | 0 | 0
subgaleal fluid collection (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 3 | 3 | 2 | 3
Confusion (Psychiatric disorders) | 3 | 2 | 1 | 3
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 2
Restlessness (Psychiatric disorders) | 1 | 0 | 0 | 0
Emotional lability (Psychiatric disorders) | 0 | 1 | 0 | 0
flat affect (Psychiatric disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
abrasion on forehead (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
cutibacterium (propionibacterium) acnes (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
erythema at site of incision (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 3 | 4 | 7
Hypotension (Vascular disorders) | 0 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT02192359/Prot_SAP_000.pdf